CLINICAL TRIAL: NCT00000601
Title: Postmenopausal Hormone Therapy in Unstable Angina
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 107; R01HL050839 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-02

CONDITIONS: Angina, Unstable; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Postmenopause
MeSH Terms: conditions — Angina, Unstable; Cardiovascular Diseases; Coronary Disease; Heart Diseases | interventions — Estrogen Replacement Therapy; Estrogens; Progesterone; Hormone Replacement Therapy

INTERVENTIONS:
Drug: estrogen replacement therapy
Drug: estrogens
Drug: progesterone
Drug: hormone replacement therapy

SUMMARY:
To determine if estrogen therapy in postmenopausal women with unstable angina reduces the incidence of ischemic episodes.

DETAILED DESCRIPTION:
BACKGROUND:

Unstable angina is a frequent diagnosis in post-menopausal women and is associated with a significant risk of myocardial infarction and need for revascularization. The pathogenesis of unstable angina involves vasoconstriction superimposed on fixed disease, causing a temporary decrease in coronary blood flow. Recent catheterization studies in patients with atherosclerosis utilizing quantitative angiography and intracoronary doppler measurements of blood flow velocity suggest that endothelial dysfunction results in a paradoxical coronary vasoconstriction response to certain neurohumoral stimuli including acetylcholine, catecholamines, and serotonin with resultant myocardial ischemia. Therapeutic agents which prevent or limit this vasoconstriction may prevent recurrent ischemia and/or myocardial infarction in unstable angina patients. Recently, estrogen receptors were identified in the smooth muscle of post-mortem human coronary arteries. Work in animal models and studies in post-menopausal women suggest that intravenous estrogen acutely decreases coronary vascular resistance, increases coronary blood flow, and prevents the paradoxical response to acetylcholine in patients with endothelial dysfunction.

DESIGN NARRATIVE:

The randomized, double-blind, placebo-controlled, multi-center trial tested the hypothesis that intravenous estrogen followed by oral estrogen and the combination of intravenous and oral estrogen and progesterone in the routine management of unstable angina were beneficial compared with placebo in post-menopausal women. Subjects with rest angina and no contraindications to hormone therapy were randomized to receive intravenous followed by oral conjugated estrogen for 21 days, intravenous estrogen followed by oral conjugated estrogen plus medroxyprogesterone for 21 days or placebo. The primary end point was the number of ambulatory electrocardiographic ischemic events over the first 48 hours. Clinical events were also determined over six months of follow-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women with unstable angina.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-07; Study Completion 2000-06 (Actual)

REFERENCES:
- [Background] Schulman SP, Thiemann DR, Ouyang P, Chandra NC, Schulman DS, Reis SE, Terrin M, Forman S, de Albuquerque CP, Bahr RD, Townsend SN, Cosgriff R, Gerstenblith G. Effects of acute hormone therapy on recurrent ischemia in postmenopausal women with unstable angina. J Am Coll Cardiol. 2002 Jan 16;39(2):231-7. doi: 10.1016/s0735-1097(01)01724-7. PMID 11788212
- [Background] Engelman RM, Pleet AB, Rousou JA, Flack JE 3rd, Deaton DW, Gregory CA, Pekow PS. What is the best perfusion temperature for coronary revascularization? J Thorac Cardiovasc Surg. 1996 Dec;112(6):1622-32; discussion 1632-3. doi: 10.1016/S0022-5223(96)70021-1. PMID 8975854